CLINICAL TRIAL: NCT00896844
Title: A Randomised Controlled Trial on the Effect of Emotional Disclosure of Traumatic Life Events on Physical Health
Brief Title: A Trial on the Effect of Emotional Disclosure of Traumatic Life Events on Physical Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Dr Catherine Meads, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Meads
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: emotional disclosure; expressive writing; students

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- emotional disclosure (Experimental): writing about emotional events from the past
  Interventions: Behavioral: emotional disclosure
- placebo writing (Placebo Comparator): writing about how they spent their time the previous day
  Interventions: Behavioral: placebo writing

INTERVENTIONS:
Behavioral: emotional disclosure — writing about emotional events from the past
  Arms: emotional disclosure
Behavioral: placebo writing — writing about how they spent their time the previous day
  Arms: placebo writing

SUMMARY:
This is a randomized, controlled trial on the effect of emotional disclosure of traumatic life events on physical health. The hypothesis is that expression of emotions could possibly improve physical health.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* any mental or physical illnesses in the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-09; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
health centre visits | within 3 months

SECONDARY OUTCOMES:
respiratory infections | within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom